CLINICAL TRIAL: NCT02679989
Title: A Randomised Controlled Trial Assessing The Impact Of An Intermittent Energy Restricted Diet On Weight Loss, Insulin Sensitivity and Heart Rate Variability In Men and Women With Central Obesity
Brief Title: The Impact Of An Intermittent Energy Restricted Diet On Insulin Sensitivity In Men and Women With Central Obesity
Acronym: Met-IER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: LighterLife (UK) Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Met-IER2016
Record Dates: First submitted 2016-01-22; First posted 2016-02-11 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2016-07

CONDITIONS: Obesity, Abdominal
Keywords: Insulin sensitivity; Weight loss; Intermittent fasting; Sympathetic nervous system
MeSH Terms: conditions — Obesity, Abdominal; Insulin Resistance; Weight Loss; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermittent Energy Restriction (Experimental): Weight loss intervention: Intermittent Energy Restriction
  Interventions: Behavioral: Intermittent Energy Restriction
- Continuous Energy Restriction (Active Comparator): Weight loss intervention: Continuous Energy Restriction
  Interventions: Behavioral: Continuous Energy Restriction

INTERVENTIONS:
Behavioral: Intermittent Energy Restriction — Dietary advice to follow 5:2 diet supported by physical activity advice and motivational group support sessions
  Arms: Intermittent Energy Restriction
Behavioral: Continuous Energy Restriction — Dietary advice to follow daily energy restricted diet supported by physical activity advice and motivational group support sessions
  Arms: Continuous Energy Restriction

SUMMARY:
An intermittent energy restricted (IER) diet may modify cardio-metabolic disease risk factors compared to an energy-matched continuous energy restricted (CER) diet. A randomised controlled parallel design trial will determine the impact of a short-term IER diet (2 consecutive days of very low calorie diet (VLCD), 5 days moderate energy restriction each week for a 4 week period), compared to a CER diet, on insulin sensitivity in healthy (disease-free) subjects with central obesity.

DETAILED DESCRIPTION:
Prediabetes rates in England have showed a marked increase, more than tripling between 2003 and 2011. It is characterised by an impaired fasting glucose or impaired glucose tolerance that increases the risk of progression to type 2 diabetes (T2D). It has been estimated that approximately 90% of T2D is attributed to excess weight. Central obesity is a primary driver of increased cardiometabolic risk due to its lipotoxicity effects, promoting a proinflammatory state that facilitates insulin resistance and beta cell dysfunction. A high waist circumference measurement, indicative of central obesity, is associated with increased risk of cardiovascular diseases and T2D, and is a stronger predictor of T2D than BMI. BMI has limitations as an indicator of adiposity since it doesn't distinguish lean from fat mass, and does not indicate body fat distribution. Conventionally, continuous energy restriction (CER) diets have been used for weight loss, which consist of a constant daily energy deficit relative to total energy expenditure. The impact on weight loss and health of an intermittent energy restriction (IER) approach has only rarely been investigated (although the "5:2 diet" has been popularised in lifestyle books aimed at the general public). An IER diet consists of a predefined period of time severely restricting energy intake, alternated with a period of greater energy intake. This approach was shown to confer metabolic benefits in overweight and obese women at risk of breast cancer with baseline BMI of 2445 (Harvie et al., 2013; Harvie et al., 2011).

Rationale: An IER diet using meal replacements (VLCD foodpacks used as total dietary replacements for 2 consecutive days each week, and a food-based energy-restricted diet for the other 5 days of the week) may modify cardio-metabolic disease risk factors compared to an energy-matched CER diet.

Research question: In centrally obese subjects, assessed by a high waist circumference measurement, does adherence to an IER diet have enhanced cardio-metabolic benefits compared to a CER diet? Hypothesis: Increases in insulin sensitivity following a 4 week dietary intervention with an IER weight loss programme will be greater compared to a standard CER programme.

Objectives:

1. A randomised controlled parallel design trial will determine the impact of a short-term IER diet compared to a CER diet on primary outcome variables (insulin sensitivity) in healthy subjects with a high waist circumference.
2. To assess the impact of an IER diet on secondary outcome variables, including body composition, heart rate variability (HRV, a measure of cardiac autonomic function, including parasympathetic and sympathetic activity), blood pressure, vascular function, other markers of insulin resistance, inflammation/adipokines, plasma lipid profile, plasma norepinephrine, ketosis, the gut microbiome and cognitive function in healthy subjects with a high waist circumference.

ELIGIBILITY:
Inclusion Criteria:

* Aged >35-75 years
* Waist circumference above cut-off for high risk of cardio-metabolic disease of >102 cm in men with a Europid, Black African and Caribbean, and other ethnic background and >88 cm in women with a Europid, Black African and Caribbean, and other ethnic background (WHO, 2008), and ≥90 cm in men and ≥80 cm in women with an Asian background (South Asian and East Asian) (Misra et al., 2009).

REFERENCES Misra A, Chowbey P, Makkar BM, Vikram NK, Wasir JS, Chadha D, et al. (2009). Consensus statement for diagnosis of obesity, abdominal obesity and the metabolic syndrome for Asian Indians and recommendations for physical activity, medical and surgical management. The Journal of the Association of Physicians of India 57: 163170.

WHO (2008). Waist circumference and waist-hip ratio: report of a WHO expert consultation. Geneva, 8-11 December 2008.

Exclusion Criteria:

* Kidney or cardiovascular disease, cancer, diabetes, gastrointestinal or chronic liver disease;
* previous bariatric surgery or other major surgery (e.g. organ transplantation);
* unable to provide written informed consent;
* have significant psychiatric disorder (e.g. schizophrenia, anxiety, panic disorder, attention deficit disorder, post-traumatic stress disorder, obsessive compulsive disorder) or uncontrolled depression;
* participated in a weight management drug trial in the previous 3 months;
* have binge eating behaviour;
* have uncontrolled epilepsy;
* alcohol or substance abuse;
* currently pregnant, lactating, or planning pregnancy within the study period;
* are using medication clinically deemed to affect metabolic rate and weight (e.g. beta blockers, corticosteroids, diuretics, etc);
* lactose intolerant.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Revised QUICKI (RQUICKI) | Baseline
  Marker of insulin sensitivity
RQUICKI | day 29
  Marker of insulin sensitivity
RQUICKI | day 31
  Marker of insulin sensitivity

SECONDARY OUTCOMES:
Plasma glucose concentration | Baseline
  Fasting
Plasma glucose concentration | day 29
  Fasting
Plasma glucose concentration | day 31
  Fasting
Plasma insulin concentration | Baseline
  Fasting
Plasma insulin concentration | day 29
  Fasting
Plasma insulin concentration | day 31
  Fasting
Plasma non-esterified fatty acid concentration | Baseline
  Fasting
Plasma non-esterified fatty acid concentration | day 29
  Fasting
Plasma non-esterified fatty acid concentration | day 31
  Fasting
Plasma total cholesterol concentration | Baseline
  Fasting
Plasma total cholesterol concentration | day 29
  Fasting
Plasma total cholesterol concentration | day 31
  Fasting
Plasma low density lipoprotein (LDL) cholesterol concentration | Baseline
  Fasting
Plasma LDL cholesterol concentration | day 29
  Fasting
Plasma LDL cholesterol concentration | day 31
  Fasting
Plasma high density lipoprotein (HDL) cholesterol concentration | Baseline
  Fasting
Plasma HDL cholesterol concentration | day 29
  Fasting
Plasma HDL cholesterol concentration | day 31
  Fasting
Plasma triglyceride concentration | Baseline
  Fasting
Plasma triglyceride concentration | day 29
  Fasting
Plasma triglyceride concentration | day 31
  Fasting
Plasma total cholesterol:HDL cholesterol ratio | Baseline
  Fasting
Plasma total cholesterol:HDL cholesterol ratio | day 29
  Fasting
Plasma total cholesterol:HDL cholesterol ratio | day 31
  Fasting
Homeostasis model assessment estimated insulin resistance (HOMA-IR) | Baseline
  Fasting (calculated from insulin and glucose)
Homeostasis model assessment estimated insulin resistance (HOMA-IR) | day 29
  Fasting (calculated from insulin and glucose)
Homeostasis model assessment estimated insulin resistance (HOMA-IR) | day 31
  Fasting (calculated from insulin and glucose)
Plasma adiponectin concentration | Baseline
  Fasting
Plasma adiponectin concentration | day 29
  Fasting
Plasma adiponectin concentration | day 31
  Fasting
Plasma leptin concentration | Baseline
  Fasting
Plasma leptin concentration | day 29
  Fasting
Plasma leptin concentration | day 31
  Fasting
Plasma interleukin-6 concentration | Baseline
  Fasting
Plasma interleukin-6 concentration | day 29
  Fasting
Plasma interleukin-6 concentration | day 31
  Fasting
Plasma beta-hydroxybutyrate concentration | Baseline
  Fasting
Plasma beta-hydroxybutyrate concentration | day 29
  Fasting
Plasma beta-hydroxybutyrate concentration | day 31
  Fasting
Plasma norepinephrine concentration | Baseline
  Fasting
Plasma norepinephrine concentration | day 29
  Fasting
Plasma norepinephrine concentration | day 31
  Fasting
Plasma soluble alpha-klotho concentration | Baseline
  Fasting
Plasma soluble alpha-klotho concentration | day 29
  Fasting
Plasma soluble alpha-klotho concentration | day 31
  Fasting
Body weight | Baseline
Body weight | day 29
Body weight | day 31
Body mass index (BMI) | Baseline
BMI | day 29
BMI | day 31
Waist circumference | Baseline
Waist circumference | day 29
Waist circumference | day 31
Hip circumference | Baseline
Hip circumference | day 29
Hip circumference | day 31
Percentage body fat | Baseline
Percentage body fat | day 29
Percentage body fat | day 31
Percentage lean body mass | Baseline
Percentage lean body mass | day 29
Percentage lean body mass | day 31
Heart rate variability (resting) | Baseline
  supine
Heart rate variability (resting) | day 29
  supine
Heart rate variability (resting) | day 31
  supine
Heart rate variability (ambulatory) | 24 h recording at baseline
Heart rate variability (ambulatory) | 24 h recording on day 29
Heart rate variability (ambulatory) | 24 h recording on day 31
Heart rate variability (sleep-time) | Baseline
Heart rate variability (sleep-time) | day 29
Heart rate variability (sleep-time) | day 31
Heart rate variability (during mental stress) | Baseline
Heart rate variability (during mental stress) | day 29
Heart rate variability (during mental stress) | day 31
Ambulatory blood pressure 24 h | 24 h analysis at baseline
Ambulatory blood pressure daytime | Daytime analysis at baseline
Ambulatory blood pressure night-time | Night-time analysis at baseline
Ambulatory blood pressure 24 h | 24 h analysis on day 29
Ambulatory blood pressure daytime | daytime analysis on day 29
Ambulatory blood pressure night-time | night-time analysis on day 29
Ambulatory blood pressure 24 h | 24 h analysis on day 31
  24 h
Ambulatory blood pressure daytime | Daytime analysis on day 31
  day time
Ambulatory blood pressure night-time | Night-time analysis on day 31
  night-time
Digital volume pulse - stiffness index (SI) | Baseline
  Stiffness index
Digital volume pulse - SI | day 29
  Stiffness index
Digital volume pulse - SI | day 31
  Stiffness index
Digital volume pulse - reflection index (RI) | Baseline
  reflection index
Digital volume pulse - RI | day 29
  reflection index
Digital volume pulse - RI | day 31
  reflection index
Mnemonic Similarity Test | Baseline
Mnemonic Similarity Test | day 29
Mnemonic Similarity Test | day 31
Power of food scale | Baseline
  questionnaire
Power of food scale | day 29
  questionnaire
Power of food scale | day 31
  questionnaire
COPE (not an acronym) | Baseline
  questionnaire
COPE | day 29
  questionnaire
COPE | day 31
  questionnaire

OTHER OUTCOMES:
Adverse events | Baseline until endpoint: day 31 (+/-1 day)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Hall, PhD, Principal Investigator — King's College London
Locations (1):
- Diabetes & Nutritional Sciences Division, King's College London, Franklin-Wilkins Buiding, 150 Stamford St., London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harvie M, Wright C, Pegington M, McMullan D, Mitchell E, Martin B, Cutler RG, Evans G, Whiteside S, Maudsley S, Camandola S, Wang R, Carlson OD, Egan JM, Mattson MP, Howell A. The effect of intermittent energy and carbohydrate restriction v. daily energy restriction on weight loss and metabolic disease risk markers in overweight women. Br J Nutr. 2013 Oct;110(8):1534-47. doi: 10.1017/S0007114513000792. Epub 2013 Apr 16. PMID 23591120
- [Background] Harvie MN, Pegington M, Mattson MP, Frystyk J, Dillon B, Evans G, Cuzick J, Jebb SA, Martin B, Cutler RG, Son TG, Maudsley S, Carlson OD, Egan JM, Flyvbjerg A, Howell A. The effects of intermittent or continuous energy restriction on weight loss and metabolic disease risk markers: a randomized trial in young overweight women. Int J Obes (Lond). 2011 May;35(5):714-27. doi: 10.1038/ijo.2010.171. Epub 2010 Oct 5. PMID 20921964
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Kim C, Pinto AM, Bordoli C, Buckner LP, Kaplan PC, Del Arenal IM, Jeffcock EJ, Hall WL, Thuret S. Energy Restriction Enhances Adult Hippocampal Neurogenesis-Associated Memory after Four Weeks in an Adult Human Population with Central Obesity; a Randomized Controlled Trial. Nutrients. 2020 Feb 28;12(3):638. doi: 10.3390/nu12030638. PMID 32121111
- [Derived] Pinto AM, Bordoli C, Buckner LP, Kim C, Kaplan PC, Del Arenal IM, Jeffcock EJ, Hall WL. Intermittent energy restriction is comparable to continuous energy restriction for cardiometabolic health in adults with central obesity: A randomized controlled trial; the Met-IER study. Clin Nutr. 2020 Jun;39(6):1753-1763. doi: 10.1016/j.clnu.2019.07.014. Epub 2019 Jul 30. PMID 31409509
- See also: Primary publication — http://www.ncbi.nlm.nih.gov/pubmed/31409509